CLINICAL TRIAL: NCT04897217
Title: Levonorgestrel-Releasing Intrauterine System (LNG-IUS) in the Management of Atypical Endometrial Hyperplasia: A Non-Inferiority Study
Brief Title: Levonorgestrel-Releasing Intrauterine System (LNG-IUS) in the Management of Atypical Endometrial Hyperplasia
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: PI decision
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00074615; WFBCCC 99321 (Other: Wake Forest Baptist Comprehensive Cancer Center); P30CA012197 (NIH)
Record Dates: First submitted 2021-05-17; First posted 2021-05-21 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-07

CONDITIONS: Endometrial Hyperplasia
MeSH Terms: conditions — Endometrial Hyperplasia | interventions — Megestrol Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Megestrol Acetate Arm - Control Arm (Active Comparator): Megestrol Acetate 160 mg by mouth daily
  Interventions: Drug: Megestrol Acetate
- Levonorgestrel IUD - Comparison Arm (Experimental): Levonorgestrel intrauterine device with 52 mg progestin (Releases 20mcg/daily)
  Interventions: Drug: Levonorgestrel Drug Implant

INTERVENTIONS:
Drug: Megestrol Acetate — The control arm will consist of oral progesterone therapy (megestrol acetate 160mg po daily). The intervention will be administered on an outpatient basis.
  Arms: Megestrol Acetate Arm - Control Arm
Drug: Levonorgestrel Drug Implant — Participants in the comparison arm will have a levonorgestrel intrauterine device placed in the office or in the operating room if the office procedure not tolerated or if they have not had a prior dilation and curettage.
  Arms: Levonorgestrel IUD - Comparison Arm

SUMMARY:
The purpose of this research study is to compare the uterus tissue of women who receive an intrauterine system to treat their endometrial hyperplasia with the uterine tissue of women who receive megestrol acetate to treat their hyperplasia. While both methods are commonly used in practice, investigators would like to see what effects each treatment has on uterine tissue.

DETAILED DESCRIPTION:
Primary Objective: To determine if Levonorgestrel-releasing intrauterine system is of equal efficacy to the standard systemic progestin therapy (megestrol acetate) based on endometrial sampling at 6 months after randomization. Non-inferiority analysis.

Secondary Objective(s):

* To determine the safety of each treatment modality.
* Determine the feasibility of transvaginal ultrasound to predict treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Complex atypical endometrial hyperplasia only. Confirmed by pathology report.
* Normal renal function and liver function tests.
* Age 18 or older.
* The effects of megestrol acetate on the developing human fetus at the recommended therapeutic dose are unknown. For this reason and because megestrol acetate is known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

Exclusion Criteria:

* Prior complex atypical endometrial hyperplasia or carcinoma.
* Prior hormone sensitive malignancy.]
* Exogenous estrogen or progestin use presently or within the past 12 months.
* Standard contraindications to progestin therapy.
* Standard contraindications to intrauterine device use.
* Simple hyperplasia, complex hyperplasia without atypia (may be present in addition to atypical endometrial hyperplasia).
* Endometrial carcinoma (worrisome or possible carcinoma not exclusionary but requires dilatation and curettage if based only on office biopsy).
* Pregnant women are excluded from this study because megestrol acetate has the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with megestrol acetate, breastfeeding should be discontinued if the mother is treated with megestrol acetate.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women of all races and ethnicity who meet the eligibility criteria are eligible for this trial. Men are excluded from participation due to the site-specific nature of the disease being studied (endometrial hyperplasia).
Enrollment: 0 (Actual)
Dates: Start 2023-06-30 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Histologic Response Scoring of Biopsy Specimens | 6 months
  The primary outcome is a response score (0: no response, 1: incomplete response, 2: complete response): Score -1 will be assigned to specimens with progression of disease (ie. Endometrial carcinoma); Score 0 will be assigned to specimens with atypical hyperplasia; Score 1 will be assigned to specimens with benign hyperplasia and will be indicative partial response to therapy; Score 2 will be assigned to specimens without hyperplasia and will be indicative of complete response to therapy. All study cases will be reviewed by a pathologist and all cases will be scored following the standard 2014 WHO classification of endometrial hyperplasia. Investigators will compare the estimated 90% confidence interval (CI) of the levonorgestrel-releasing Intrauterine system versus the standard therapy from the noninferiority trial to a predefined margin.

SECONDARY OUTCOMES:
Number of Toxicities for Each Treatment | Up to 8 months
  Toxicities for each treatment modality based on standard toxicity scoring using NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Investigators will compare the number of toxicities between the two treatment groups using chi-squared tests.
Pathological Response to Treatment | Up to 8 months
  The pathological response variable will be treated as a binary variable, the Wilcoxon rank sum test will be used to explore the association between measurement of the endometrial stripe and the response outcome at each visit. Score -1 will be assigned to specimens with progression of disease (ie. Endometrial carcinoma); Score 0 will be assigned to specimens with atypical hyperplasia; Score 1 will be assigned to specimens with benign hyperplasia and will be indicative partial response to therapy; Score 2 will be assigned to specimens without hyperplasia and will be indicative of complete response to therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Janelle Darby, MD, Principal Investigator — Wake Forest Baptist Health Sciences

IPD SHARING:
Plan to Share IPD: No